CLINICAL TRIAL: NCT05569915
Title: Project QueST 2023: Queer Survivors of Trauma
Acronym: QueST2023
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: Yale University (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jillian Scheer, Assistant Professor, Cobb-Jones Professor Clinical Psychology, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-306
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Stress Disorders, Post-Traumatic; Drinking Heavy
Keywords: sexual trauma; PTSD symptoms; coping; LGBTQ; lesbian; bisexual; Sexual and Gender Minorities; Alcohol-Related Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sexual Trauma; Homosexuality, Female; Bisexuality; Coitus; Alcohol-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trauma Expressive Writing (Experimental): In the trauma condition, we ask participants to write about a traumatic experience, prompting them to write their very deepest thoughts and feelings about the most traumatic experience of their entire life or an extremely important stressful, upsetting, or emotional issue that has affected them.
  Interventions: Behavioral: Trauma Expressive Writing
- Stigma Expressive Writing (Experimental): In the stigma condition, we ask participants to write about an experience of stigma, prompting them to write about their very deepest thoughts and feelings about the most difficult or painful experience of stigma or bias (e.g., prejudice, bullying, rejection, discrimination) based on one or more of their identities (e.g., race/ethnicity, gender identity, sexual identity, religion) that they have faced.
  Interventions: Behavioral: Stigma Expressive Writing
- Control (Placebo Comparator): In the control condition, we ask participants to write about their day, prompting them to write about what they did yesterday from the time they got up until the time they went to bed.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Trauma Expressive Writing — Participants assigned to the trauma condition will write about an experience of trauma for 15 to 20 minutes per day across five consecutive days.
  Arms: Trauma Expressive Writing
Behavioral: Stigma Expressive Writing — Participants assigned to the stigma condition will write about an experience of stigma or bias for 15 to 20 minutes per day across five consecutive days.
  Arms: Stigma Expressive Writing
Behavioral: Control — Participants assigned to the control condition will write about their days for 15 to 20 minutes per day across five consecutive days. This control condition is standard across many expressive writing studies.
  Arms: Control

SUMMARY:
This study aims to test the initial efficacy of tailored online writing interventions specifically designed for sexual minority women, transgender individuals, and/or nonbinary people to target the primary outcomes: posttraumatic stress disorder (PTSD) symptom severity and hazardous drinking.

DETAILED DESCRIPTION:
This study aims to provide a novel method for adapting and testing evidence-based expressive writing (EW) treatments for trauma-exposed sexual minority women (SMW) and gender diverse individuals. The investigators will (1) describe the development and components of the proposed EW treatments, (2) discuss our plan for evaluating acceptability and feasibility of the proposed study, (3) identify steps for characterizing preliminary efficacy of EW treatments in reducing PTSD symptom severity and hazardous drinking levels compared to control, and (4) highlight our strategy for preliminarily evaluating mediators and moderators of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* being at least 18 years of age
* reporting English fluency
* identifying as sexual minority women, inclusive of gender-diverse people
* living in the United States (US)
* reporting one or more Criterion A traumatic events
* having internet and email access
* not having received inpatient psychiatric support in the past six months

Exclusion Criteria:

* failing an inclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women who are assigned female at birth, transgender men or women, and nonbinary people regardless of sex assigned at birth.
Enrollment: 131 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptom severity | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Posttraumatic stress disorder (PTSD) symptoms will be measured with the Psychometric Properties of the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5). The PDS-5 is a 24-item self-report measure designed to assess the severity of DSM-5 PTSD symptoms. The 24-item scale comprises a checklist of traumatic event types the individual has experienced, identification of the most distressing traumatic event, and an assessment of PTSD symptoms. The assessment of PTSD symptoms yields a total score and three subscales (re-experiencing, avoidance, and arousal), and a cutoff score of 28 or higher indicates a probable PTSD diagnosis. Items are scored 1 = once a week or less/a little to 4 = 6 or more times a week/severe. At baseline and 3-month follow-up assessments, participants will complete the PDS-5 in reference to the past month. At the one-week follow-up assessment, participants will complete the PDS-5 in reference to the past week.
Change in hazardous drinking levels | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  The Alcohol Use Disorders Identification Test (AUDIT) will be used to measure hazardous drinking levels. The AUDIT is a 10-item screening measure of problematic alcohol use with individual items ranging from 0 to 4. Scores of 8 and higher are thought to reflect hazardous alcohol use. At baseline and 3-month follow-up assessments, participants will complete the AUDIT in reference to the past month.
Change in drinking quantity | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  To assess drinking quantity in the past week, the investigators will ask participants one question that assesses retrospective estimates for number of drinks consumed on average (in a typical week). The investigators will assess change in the total number of drinks consumed on a typical week in the past month from baseline to total number of drinks consumed in the past week at one-week follow-up and from baseline to total number of drinks consumed in a typical week in the past month at 3-months follow-up assessment. At baseline and 3-month follow-up assessments, participants will complete the hazardous drinking quantity question in reference to a typical week during the past month. At the one-week follow-up assessment, participants will complete the hazardous drinking quantity question in reference to the past week.
Change in heavy drinking frequency | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  The investigators will assess the number of heavy drinking days (days where participants assigned female or intersex at birth consume ≥4 standard drinks and participants assigned male at birth consume ≥5 standard drinks). Response options range from 0 = never to 4 = almost every day where higher scores represent greater heavy drinking frequency. The investigators will assess change in frequency of heavy drinking days in the past month from baseline to frequency of heavy drinking days in the past week at one-week follow-up and from baseline to frequency of heavy drinking days in the past month at 3-months follow-up. At baseline and 3-month follow-up assessments, participants will report frequency of heavy drinking days over the past month. At the one-week follow-up assessment, participants will report frequency of heavy drinking days over the past week.

SECONDARY OUTCOMES:
Change in trauma centrality. | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Trauma centrality will be measured with the Centrality of Events Scale (CSE), which assesses to what degree an event is integrated into an individual's life story and identity. The 20-item questionnaire represents three factors of which the memory of the event has become an (a) reference point for everyday inferences, (b) a core part of personal identity, and (c) a turning point in the life story. Items are rated on a scale from 1 (totally disagree) to 5 (totally agree), and summed to yield a total score.
Change in coping. | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Coping will be measured using the Brief COPE, a 28-item measure that assesses coping strategies during stress. The Brief COPE consists of 14 subscales with two items per subscale. The investigators will use eight items across four subscales: self-distraction, denial, behavioral disengagement, and self-blame. Respondents rate items using a four-point Likert scale ranging from 1 ("I haven't been doing this at all") to 4 ("I've been doing this a lot"). Greater scores indicate greater use of self-distraction, denial, behavioral disengagement, and self-blame to cope with stress.
Change in sexual minority identity-related experiences | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Sexual minority identity-related experiences will be assessed with the Lesbian, Gay, Bisexual Identity Scale. This scale contains 27 items and assesses concealment, internalized stigma, and anticipated stigma, among other identity-related constructs. Responses range from 1 (Disagree strongly) to 6 (Agree strongly). Subscale scores are computed by reverse-scoring items as needed and averaging subscale item ratings. Subscale composition is as follows: Acceptance Concerns (5, 9, 16), Concealment Motivation (1, 4, 19), Identity Uncertainty (3, 8, 14, 22), Internalized Homonegativity (2, 20, 27), Difficult Process (12, 17, 23), Identity Superiority (7, 10, 18), Identity Affirmation (6, 13, 26), and Identity Centrality (11, 15, 21, 24, 25).
Change in perceived stress. | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Perceived stress will be measured with the Ten-Item Perceived Stress Scale (PSS-10), a 10-item self-reporting measure to assess the level of stress experienced by the respondents. Items are scored on a five-point Likert scale, from 0 (never) to 4 (very often). Greater scores indicate greater perceived stress. At baseline and 3-month follow-up assessments, participants will complete the PSS-10 in reference to the past month. At the one-week follow-up assessment, participants will complete the PSS-10 in reference to the past week.
Change in depression and anxiety symptoms. | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Depression and anxiety symptoms will be assessed using the Brief Symptom Inventory (BSI). The BSI uses 18 items across 2 subscales to capture the extent to which an individual has been distressed by various symptoms of depression and anxiety over the past week (e.g., "Nervousness or shakiness inside" for the anxiety subscale and "Feeling hopeless about the future" for the depression subscale). Possible response options range from 0 (Not at all) to 4 (Extremely). Greater scores indicate greater depression and anxiety symptom severity. At baseline, 1-week, and 3-month follow-up assessments, participants will complete the depression and anxiety subscales in reference to the past week.
Change in emotion regulation. | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Emotion regulation will be assessed with the Difficulties in Emotion Regulation Scale (DERS). The Difficulties in Emotion Regulation Scale contains 36 items that capture the extent to which an individual generally has trouble regulating their emotions. The investigators will use the distress tolerance and ability to tolerate negative emotions subscales. Possible responses range from 1 (Almost never; 0-10% of the time) to 5 (Almost always; 91-100% of the time). Greater total scores indicate greater difficulties with emotion regulation (i.e., emotion dysregulation).
Change in impulsivity. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Impulsivity will be measured with the Short UPPS-P, a 20-item, self-report questionnaire that measures five dimensions of impulsive behavior (negative urgency, lack of premeditation, lack of perseveration, sensation seeking, and positive urgency). Each item is rated on a 4-point scale, from Agree strongly (1) to Disagree strongly (4). The investigators will use the negative urgency subscale from the UPPS-P. Items are reverse scored such that higher scores indicate greater negative urgency (i.e., impulsivity).
Change in self-efficacy. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Self-efficacy will be measured by the Generalized Self-Efficacy Scale (GSES). The GSES is a measure of general self-efficacy. It consists of 10 items. Respondents rate each item on a 1 (not true at all) to 4 (exactly true) scale. Higher scores represent greater self-efficacy.
Change in attachment style. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Attachment style will be measured using the Experiences in Close Relationships - Short form (ECR- SF). The investigators will use the 6-item anxiety subscale and 6-item avoidance subscale. The ECR uses a 6-point scale to assess both anxious attachment and avoidant attachment. Response options range from 1 = strongly disagree to 6 = strongly agree where higher scores represent greater anxiety and avoidant attachment styles.
Change in self-compassion. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Self-compassion will be measured with the Self-Compassion Scale (SCS), a 26-item self-report measure of the degree to which individuals exhibit a kind and accepting attitude toward themselves. The investigators will use the following subscales of the SCS: self-kindness, common humanity, and mindfulness. Responses are on a Likert-type scale from 1 = almost never to 5 = almost always, with higher scores indicating greater self-compassion.
Change in suicidality. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Suicidality will be measured with the SBQ-R. Suicide ideation/behavior will be assessed using Item 1 of the SBQ-R. The original SBQ-R consists of four items but only the aforementioned item was used in the current study due to space constraints. However, Item 1 of the SBQ-R has been recommended for screening purposes and has repeatedly been used in clinical and non-clinical samples. Response options range from 0 = Never to 5 = I have attempted to kill myself, and really hoped to die. At baseline and 3-month follow-up assessments, participants will complete the SBQ-R in reference to the past 3 months.
Change in hope. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Hope was measured with a hope scale - a single question. Participants will rate their answers on a visual analog scale from 1 ("not at all hopeful") to 10 ("very hopeful"). Higher scores represent greater hope.
Change in substance use. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Substance use will be assessed using the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), a screening measure of severity of involvement using alcohol, cannabis, cocaine, prescription stimulants, amphetamine-type stimulants, sedatives and sleeping pills, hallucinogens, inhalants, street opioids, prescription opioids, and other miscellaneous drugs. Response options include 0 = no, 1 = yes, but not in the past 3 months, and 2 = yes, in the past 3 months. At baseline and 3-month follow-up assessments, participants will complete the ASSIST in reference to past 3 months use.
Change in problematic drug use. | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Problematic drug use will be measured with the Drug Use Disorders Identification Test (DUDIT). The DUDIT is a self-report instrument composed of 11 items identifying problems related to substance use. Scoring of the DUDIT is two-fold: items 1 to 9 are scored on a five-point Likert scale, while items 10 and 11 are scored on a three-point scale. The overall score is calculated by summing the scores on all items. Higher scores represent greater problematic drug use. At baseline and 3-month follow-up assessments, participants will complete the DUDIT in reference to past 3 months use.
Change in heavy drinking presence | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Heavy drinking presence will be measured by asking if participants had 4 of more drinks if assigned female at birth or intersex OR 5 or more drinks if assigned male at birth in the past 3 months. At baseline and 3-month follow-up assessments, participants will answer the question about heavy drinking presence in reference to past 3 months.
Change in alexithymia | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Alexithymia will be measured with the Perth Alexithymia Questionnaire (4-item negative-difficulty identifying feelings subscale and 4-item negative-difficulty describing feelings subscale). The Perth Alexithymia Questionnaire (PAQ) is a 24-item self-report measure of alexithymia answered on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). Subscales can be summed to derive an overall alexithymia total score, with higher scores indicative of higher levels of alexithymia.
Change in dissociation | Baseline (Pre-intervention), Immediate Post-intervention (1 week post first treatment session), and Three-month Follow-up (3 months post first treatment session)
  Dissociation will be measured with the Brief Dissociative Experiences Scale (DES-B) - Modified, which was recently Modified for DSM-5. The DES-B is an eight items scale that measures the phenomena of dissociative experience over the past week, not necessarily pathological dissociation. Response options range from 0 to 4, with 0 indicating not at all, and 4 more than once a day. At baseline, 1-week, and 3-month follow-up assessments, participants will complete the DES-B in reference to the past week.
Change in general health perceptions | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  Physical health symptoms will be assessed using the first item of the Short-Form Health Survey (SF-12). Response options are on a 5-point Likert-scale with higher scores indicating worse general health perceptions. Scores range from Excellent (0) to Poor (4).
Change in physical health symptoms | Baseline (Pre-intervention) and Three-month Follow-up (3 months post first treatment session)
  The investigators will also assess physical health symptoms using the Patient Health Questionnaire - 15 (PHQ-15), a self-administered somatic symptoms subscale derived from the full PHQ. Participants are asked to rate the severity of their symptoms during the previous 4 weeks on a 3-point scale as either 0 ("not bothered at all"), 1 ("bothered a little") or 2 ("bothered a lot"). Total symptom severity score ranged from 0 to 30. At baseline and 3-month follow-up assessments, participants will answer the questions about physical health symptoms in reference to the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian R Scheer, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion for three years.
Access Criteria: Data access requests from qualified academic investigators for non-commercial research interests will be reviewed by study investigators. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] World Health Organization, Babor, Thomas F., Higgins-Biddle, John C., Saunders, John B. Monteiro, Maristela G. AUDIT: The Alcohol Use Disorders Identification Test: Guidelines for use in primary health care, 2nd ed. World Health Organization. 2001. https://apps.who.int/iris/handle/10665/67205
- [Background] Dalenberg C, Carlson E. New versions of the Dissociative Experiences Scale: The DES-R (revised) and the DES-B (brief). Paper presented at the International Society for Traumatic Stress Studies Annual Meeting. 2010;26:203. https://istss.org/meetings-events/meeting-archives/2010-annual-meeting-archives.aspx
- [Background] Preece D, Becerra R, Robinson K, Dandy J, Allan A. The psychometric assessment of alexithymia: Development and validation of the Perth Alexithymia Questionnaire. Pers Individ Dif. 2018;132:32-44. doi: 10.1016/j.paid.2018.05.011
- [Background] Salomon K, Bosson JK, El-Hout M, Kiebel E, Kuchynka SL, Shepard SL. The Experiences with Ambivalent Sexism Inventory (EASI). Basic Appl Soc Psychol. 2020;42(4):235-253. doi: 10.1080/01973533.2020.1747467
- [Background] Tebbe EA, Moradi B, Wilson E, Bell HL, Connelly K, Lenzen A. Development and psychometric evaluation of the Sexual Minority Women's Sexual Objectification Experiences Scale. J Couns Psychol. 2021 Oct;68(5):501-514. doi: 10.1037/cou0000547. Epub 2021 Mar 25. PMID 33764114
- [Background] Gomez JM. What's the harm? Internalized prejudice and cultural betrayal trauma in ethnic minorities. Am J Orthopsychiatry. 2019;89(2):237-247. doi: 10.1037/ort0000367. Epub 2018 Nov 8. PMID 30407029
- [Background] Hildebrand M. The Psychometric Properties of the Drug Use Disorders Identification Test (DUDIT): A Review of Recent Research. J Subst Abuse Treat. 2015 Jun;53:52-9. doi: 10.1016/j.jsat.2015.01.008. Epub 2015 Jan 31. PMID 25682718
- [Background] Carter G, Yu Z, Aryana Bryan M, Brown JL, Winhusen T, Cochran G. Validation of the tobacco, alcohol, prescription medication, and other substance use (TAPS) tool with the WHO alcohol, smoking, and substance Involvement screening test (ASSIST). Addict Behav. 2022 Mar;126:107178. doi: 10.1016/j.addbeh.2021.107178. Epub 2021 Nov 10. PMID 34802777
- [Background] Berntsen D, Rubin DC. The centrality of event scale: a measure of integrating a trauma into one's identity and its relation to post-traumatic stress disorder symptoms. Behav Res Ther. 2006 Feb;44(2):219-31. doi: 10.1016/j.brat.2005.01.009. PMID 16389062
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Neff, K. D. (2003). Development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250.
- [Background] Osman A, Bagge CL, Gutierrez PM, Konick LC, Kopper BA, Barrios FX. The Suicidal Behaviors Questionnaire-Revised (SBQ-R): validation with clinical and nonclinical samples. Assessment. 2001 Dec;8(4):443-54. doi: 10.1177/107319110100800409. PMID 11785588
- [Background] Gandhi SK, Salmon JW, Zhao SZ, Lambert BL, Gore PR, Conrad K. Psychometric evaluation of the 12-item short-form health survey (SF-12) in osteoarthritis and rheumatoid arthritis clinical trials. Clin Ther. 2001 Jul;23(7):1080-98. doi: 10.1016/s0149-2918(01)80093-x. PMID 11519772
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Mohr JJ, Kendra MS. Revision and extension of a multidimensional measure of sexual minority identity: the Lesbian, Gay, and Bisexual Identity Scale. J Couns Psychol. 2011 Apr;58(2):234-245. doi: 10.1037/a0022858. PMID 21319899
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of psychopathology and behavioral assessment, 26(1), 41-54.
- [Background] Verdejo-Garcia A, Lozano O, Moya M, Alcazar MA, Perez-Garcia M. Psychometric properties of a Spanish version of the UPPS-P impulsive behavior scale: reliability, validity and association with trait and cognitive impulsivity. J Pers Assess. 2010 Jan;92(1):70-7. doi: 10.1080/00223890903382369. PMID 20013458
- [Background] Luszczynska A, Scholz U, Schwarzer R. The general self-efficacy scale: multicultural validation studies. J Psychol. 2005 Sep;139(5):439-57. doi: 10.3200/JRLP.139.5.439-457. PMID 16285214
- [Background] Wei M, Russell DW, Mallinckrodt B, Vogel DL. The Experiences in Close Relationship Scale (ECR)-short form: reliability, validity, and factor structure. J Pers Assess. 2007 Apr;88(2):187-204. doi: 10.1080/00223890701268041. PMID 17437384
- [Result] Foa EB, McLean CP, Zang Y, Zhong J, Powers MB, Kauffman BY, Rauch S, Porter K, Knowles K. Psychometric properties of the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5). Psychol Assess. 2016 Oct;28(10):1166-1171. doi: 10.1037/pas0000258. Epub 2015 Dec 21. PMID 26691504